CLINICAL TRIAL: NCT04117828
Title: Assessment of Glycemic Index of Different Dates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, NASEER AHMED, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NA124
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Glycemic Index and Glycemic Load
MeSH Terms: interventions — Chronology as Topic

STUDY DESIGN:
Intervention Model Description: 40 participants will be included in the study and will be divided into four groups. The AKU faculty and staff will be invited to MDL with fasting of 12 hr. Written informed consent (a copy will also be provided to the participant) will be taken from each individual.Following vitals will be measured body weight, height and blood pressure. 1st group will be the control that will consume 50 g of glucose and 2nd, 3rd, and 4th group will consume 50 g of different kinds of dates. Their blood sugar level will be checked at 0, 30, 60, 90 and 120 mins. Glycemic index and glycemic load will be calculated and will be compared.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): 50 g of glucose will be given to the individuals
  Interventions: Dietary Supplement: Dates
- 1st Intervention group (Experimental): 50 g of Aseel dates will be given to the individuals
  Interventions: Dietary Supplement: Dates
- 2nd Intervention group (Experimental): 50 g of Ajwa dates will be given to the individuals
  Interventions: Dietary Supplement: Dates
- 3rd Intervention group (Experimental): 50 g of Karbala dates will be given to the individuals
  Interventions: Dietary Supplement: Dates

INTERVENTIONS:
Dietary Supplement: Dates — Phoenix dactylifera, commonly known as date or date palm is a flowering plant species in the palm family, Arecaceae. Dates are the fruit of the date palm tree, which is grown in many tropical regions of the world. Dates provide a wide range of essential nutrients, and has certain protective effects on health of individuals.

SUMMARY:
Glycemic Index is a system of classification of different foods with significant levels of carbohydrates based on how they affect blood glucose levels after being consumed. In this study we will compare glycemic index of different varieties

DETAILED DESCRIPTION:
Glycemic Index is a system of classification of different foods with significant levels of carbohydrates based on how they affect blood glucose levels after being consumed. Despite being a significant parameter of blood glucose, GI does not depict the effect of the food when taken in a controlled recommended amount, and so the Glycemic Loads (GL) must also be calculated, thereby measuring the impact on glycemic levels after consumption of standard food portion sizes. Dates are high energy foods consumed in various parts of the world, are known to be a source of several important nutrients and are also shown to have significant impacts in preventing illnesses due to their anti-inflammatory and anti-microbial actions as well as preventative action against oxidative reactions The greatly frequent consumption of dates necessitates the identification of their GI and GL to ensure whether consumption is beneficial and safe for individuals. The objective of the study is to determine and compare the values of GI and GL of three varieties of dates in order to assess their safe consumption by individuals

ELIGIBILITY:
Inclusion Criteria:

* General population from AKU
* Adult ages (18- 60 years) will be included in the study

Exclusion Criteria:

* Individuals with Dates/Ajwa allergy
* Pregnant women and individuals with diabetes, metabolic syndrome or any other co-morbidity will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose level | 1 week
  Estimation of glycemic index and glycemic load

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Ahmed, Ph.D, Principal Investigator — AKU
Locations (1):
- Agha Khan University Hospital, Karachi, Sindh, Pakistan